CLINICAL TRIAL: NCT02304874
Title: Evaluation of Body Iron Stores in Overweight Healthy Volunteers
Acronym: FERNORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOC/11-03
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers; Overweight
Keywords: Ferritins; Iron Overload; Metabolic Syndrome; Venesection therapy; Volunteers
MeSH Terms: conditions — Overweight; Iron Overload; Metabolic Syndrome | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phlebotomy (Other): Phlebotomies will be performed every 14 days at the Clinical Investigation Unit (CIU) until the value of ferritin level is below 50 µg/mL and/or the value of hemoglobin level is below 12 g/dL.
  Interventions: Other: Phlebotomy

INTERVENTIONS:
Other: Phlebotomy

SUMMARY:
Normal body iron store value in overweight subjects is currently not described in literature. The comparison of this value with body iron levels in patients suffering from dysmetabolic iron overload syndrome (DIOS) could allow to quantify iron overload in this condition. The purpose of the study is to determine iron levels in healthy overweight volunteers, and to compare them to DIOS patients treated with phlebotomy.

DETAILED DESCRIPTION:
Normal body iron store value in overweight subjects is currently not described in literature. The comparison of this value with body iron levels in patients suffering from dysmetabolic iron overload syndrome (DIOS) could allow to quantify iron overload in this condition.

DIOS is the leading cause of hyperferritinemia and mainly affects men between 45 and 60 years. It is characterized by unexplained hyperferritinemia associated to metabolic disorders (including overweight) and iron overload, objectified by MRI or liver biopsy.

Some authors suggest that hyperferritinemia associated to metabolic disorders is the expression of an inflammatory syndrome caused by insulin resistance and steatohepatitis, and not the manifestation of real iron overload.

The debate surrounding iron overload in DIOS is related to the limits of the current analysis methods (phlebotomy, liver iron concentration, MRI). At present, phlebotomy is the standard method used to determine body iron stores.

Using this method, the purpose of the study is to determine iron levels in healthy overweight volunteers, and to compare them to DIOS patients treated with phlebotomy included in another ongoing clinical trial (SAIGNEES - ClinicalTrials.gov Identifier: NCT01045525).

ELIGIBILITY:
Inclusion Criteria:

* Male,
* At least 18 years old
* BMI > 25 Kg/m2
* Serum ferritin level between 100 et 300 µg/L
* Written informed consent

Exclusion Criteria:

* Blood donations in the past two years
* Alcohol consumption more than 30 g/day
* Inflammatory syndrome (CRP > 10 mg/L)
* Inflammatory, dysimmunitary or cancerous disease
* Hepatic cytolysis
* Transferrin saturation > 45%
* Person involved in another clinical trial
* Person with a measure of legal protection (guardianship)
* Person who reached the annual limit for compensation provided by biomedical research
* Hemoglobin < 13 g/dL
* Uncontrolled heart failure or coronary insufficiency
* Abnormal ECG
* Echocardiographic abnormalities contraindicating phlebotomy
* Hepatic, renal or respiratory insufficiency
* Superficial venous network insufficiency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Amount of mobilized iron (AMI) in grams collected by phlebotomies to have a ferritin level < 50 µg/L | Every 14 days, up to 3 months
  Phlebotomies will be performed every 14 days at the Clinical Investigation Unit, until ferritin level is below 50 µg/mL and/or hemoglobin is below 12 g/dL.

SECONDARY OUTCOMES:
Serum hepcidin level variation during the phlebotomy | Every 14 days, up to 3 months
Serum soluble transferrin receptor variation during the phlebotomy | Every 14 days, up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Laviolle, MD, PhD, Study Chair — Centre d'Investigation Clinique Inserm 1414, Service de Pharmacologie Clinique, Hôpital de Pontchaillou; Caroline Jezequel, MD, Principal Investigator — Centre d'Investigation Clinique Inserm 1414, Service de Pharmacologie Clinique, Hôpital de Pontchaillou
Locations (1):
- CHU Pontchaillou, Rennes, France

REFERENCES:
- [Result] Jezequel C, Laine F, Laviolle B, Kiani A, Bardou-Jacquet E, Deugnier Y. Both hepatic and body iron stores are increased in dysmetabolic iron overload syndrome. A case-control study. PLoS One. 2015 Jun 1;10(6):e0128530. doi: 10.1371/journal.pone.0128530. eCollection 2015. PMID 26030828